CLINICAL TRIAL: NCT05145634
Title: The Effectiveness of Interactive Nursing Education Program Through Health Belief Model Based and Informative Technology-assisted on Atrial Fibrillation Patients Receiving Oral Anticoagulant: A Randomized Control Trial
Brief Title: The Effectiveness of Interactive Nursing Education Program Through Health Belief Model Based and Informative Technology-assisted on Atrial Fibrillation Patients Receiving Oral Anticoagulant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 103-5623B
Record Dates: First submitted 2021-07-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation
Keywords: health education program; health belief model; informative technology; anticoagulants; atrial fibrillation; randomized controlled study
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational group (Experimental): The interventions administered to the experimental group were one-on-one instruction and Health Brief Model (HBM)-driven strategies, health information technology system, monthly telephone follow-ups, and providing medication cards.
  Interventions: Other: Patient education related oral anticoagulants (OACs)
- Control group (No Intervention): Patients in the control group only received brochure and medication cards.

INTERVENTIONS:
Other: Patient education related oral anticoagulants (OACs) — The interventions administered to the experimental group were one-on-one instruction and Health Belief Model (HBM)-driven strategies, health information technology system, monthly telephone follow-ups, and providing medication cards. Patient education related oral anticoagulant: each subject in the experimental group was taught individually according to investigators' App in the outpatient department (OPD) by researchers. Every months, participants received a follow-up phone call to clarify any questions related to the knowledge of anticoagulants. The contents of the teaching material consisted of: the purpose of taking anticoagulant, side effects, adjustments to daily diet, and precautions (i.e.how to take medication safely, interaction between foods and medicine, prevention and checking of signs and symptoms of bleeding). The control group received the brochure and medical card after pretest and routine care in the OPD. All participants completed posttest at 3-month follow-up.
  Arms: Educational group

SUMMARY:
This study examined patients on taking oral anticoagulants (OACs) are often prescribed for Atrial fibrillation (AFib) to determine the effectiveness of a multiple interactive health education program, which was developed based on the health belief model (HBM) and incorporated information technologies.

DETAILED DESCRIPTION:
A randomized controlled study was conducted on the cardiology outpatients. The patients were recruited through purposive sampling. The participants had been diagnosed with AFib and were receiving OACs. The participants were divided according to the blocks of clinic hours and assigned randomly to the experimental group or control group. The control variables involved demographic characteristics and medical history. The dependent variables and corresponding research instruments were medication knowledge and health beliefs, medication satisfaction and quality of life (QoL). Other than the medication knowledge questionnaire, which was assessed monthly, all the measurement instruments were applied twice: first in a pretest, and again in a posttest administered at the third month. The interventions administered to the experimental group were one-on-one instruction and HBM-driven strategies, health information technology system, monthly telephone follow-ups, and providing medication cards. The participants in the control group only received brochure and medication cards.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Atrial Fibration by a physician and taking oral anticoagulant as treatment
* 20years old or older
* clear consciousness for communication
* willingness to participate in research.

Exclusion Criteria:

* can not communicate clearly
* without willingness to participate in research

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The change of "medication knowledge of anticoagulants" | medication knowledge of anticoagulants was assessed at baseline, change from baseline medication knowledge of anticoagulants at 2 months, and change from baseline medication knowledge of anticoagulants at 3 months
  There were 11 questions related to knowledge of anticoagulants designed by investigators' research team. The range of scores was 0-22. The higher the score, the better the participants' knowledge of anticoagulants was.
The change of "health beliefs of anticoagulants" | health beliefs of anticoagulants were assessed at baseline, and change from baseline health beliefs of anticoagulants at 3 months
  There were 22 questions related to health beliefs of anticoagulants designed by investigators' research team. The range of scores was 0-88. The higher the score, the better the participants' health beliefs was.

SECONDARY OUTCOMES:
The change of "medication satisfaction of anticoagulants" | medication satisfaction of anticoagulants was assessed at baseline, and change from baseline medication satisfaction of anticoagulants at 3 months
  There were 26 questions related to medication satisfaction of anticoagulants (Duke Anticoagulation Satisfaction Scale, DASS). The range of scores was 1-182. The lower the score, the better the participants' medication satisfaction was.
The change of "quality of life for patients taking anticoagulants" | quality of life for patients taking anticoagulants was assessed at baseline, and change from baseline quality of life for patients taking anticoagulants at 3 months
  There were 12 questions related to quality of life for patients taking anticoagulants (Short Form-12, SF-12). The range of scores was 0-100 transferred in each question. The higher the score, the better the participants' quality of life was.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsia Tsai, Principal Investigator — Chang Gung University

REFERENCES:
- [Background] Konieczynska, M., Sobieraj, E., Bryk, A. H., Debski, M., Polak, M., Podolec, P., . . . Undas, A. (2018). Differences in knowledge among patients with atrial fibrillation receiving NOACs and vitamin K antagonists. Kardiol Pol. doi:10.5603/KP.a2018.0069 Morrissey, E. C., Casey, M., Glynn, L. G., Walsh, J. C., & Molloy, G. J. (2018). Smartphone apps for improving medication adherence in hypertension: patients' perspectives. Patient Prefer Adherence, 12, 813-822. Stephenson, J. J., Shinde, M. U., Kwong, W. J., Fu, A. C., Tan, H., & Weintraub, W. S. (2018). Comparison of claims vs patient-reported adherence measures and associated outcomes among patients with nonvalvular atrial fibrillation using oral anticoagulant therapy. Patient Prefer Adherence, 12, 105-117.